CLINICAL TRIAL: NCT03576222
Title: Prospective, Randomized, Comparative Study About Effects of Preventive Negative Pressure Therapy With PICO or Standard Care Dressing (MEPORE) on Surgical Wounds After Large Incisional Hernia Repair
Brief Title: Preventive PICO on Surgical Wounds After Large Incisional Hernia Repair
Acronym: PICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, JOSE BUENO-LLEDÓ, HEAD OF SECTION, Hospital Universitario La Fe
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PICO-01
Record Dates: First submitted 2018-06-09; First posted 2018-07-03 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Incisional Hernia
Keywords: PICO; incisional hernia; surgical site occurrences
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Intervention Model Description: PICO dressing prevents surgical site ocurrences after abdominal Wall repair
Who Masked: Participant
Masking Description: intraoperative use of randomized dressing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with preventive PICO (Active Comparator): PICO dressing is used in patients with incisional hernia intraoperatively
  Interventions: Device: PICO DRESSING
- patients with preventive MEPORE (Placebo Comparator): MEPORE dressing is used in patients with incisional hernia intraoperatively
  Interventions: Device: MEPORE dressing

INTERVENTIONS:
Device: PICO DRESSING — USE PICO DRESSING ON SURGICAL INCISION AFTER ABDOMINAL WALL REPAIR IN THE SURGICAL ROOM
  Arms: patients with preventive PICO
Device: MEPORE dressing — MEPORE dressing
  Arms: patients with preventive MEPORE

SUMMARY:
To determine the efficacy on decreasing the rate of surgical wound complications in patients undergoing repair of large incisional hernias, after the prophylactic application of a single-use negative pressure therapy dressing (PICO), versus a conventional dressing.

DETAILED DESCRIPTION:
Hypothesis The preventive use of single-use PICO dressing reduces the complications of the surgical wound (infection and dehiscence of the surgical wound) in patients after large incisional hernia repair.

Objectives

Primary:

To determine the efficacy on decreasing the rate of surgical wound complications in patients undergoing eventration surgery, after the prophylactic application of a single-use negative pressure therapy (NPT) dressing, as opposed to a conventional dressing.

Secondary:

* To report the incidence of wound infection and dehiscence during the patient's admission, at 7 days, 15 days and month after surgical repair applying a conventional dressing (MEPORE) or PICO dressing.
* To quantify economic costs applying a PICO dressing versus a MEPORE dressing.

Methods:

Selection of patients Collection of the sample will be made in the Abdominal Wall Surgery Unit (La Fe Hospital), according to the inclusion and exclusion criteria. The surgeon will explain to the patient the objectives of the study and will give him an informed consent and will answer all the doubts about the study.

Patients will be assigned to two groups in a 1: 1 ratio. Assignment of each patient to the different groups will be done using a randomized method according to the following distribution:

* Group A, it will be applied the dressing object of study (PICO)
* Group B, it will be applied the conventional dressing (MEPORE).

Data collection and Study variables

For each patient, the data collection notebook designed for this purpose must be completed, which includes the following study variables:

1. Dependent (study outcomes)

   * Infection and dehiscence of surgical wound. These variables will be assessed throughout the admission and at 7 and 30 days from the hernia repair, during hospital stay, and at 15 days in the Unit.
   * Variables related to direct costs (hospital stay, material, antibiotic use, operating room use, etc). Other variables related to indirect costs (time of cure by nursing).
2. Independent

   * Demographic data: age, sex, BMI.
   * Classification ASA (American Society of Anesthesiologists)
   * Risk factors abour surgical wound complications: drainage, preoperative chemotherapy, preoperative radiotherapy, Diabetes Mellitus, cardiovascular disease, immunosuppressive treatment, active smoking, obesity, hypertension, inflammatory bowel disease.

Number of subjects 150 patients undergoing hernia repair of large incisional hernia (types W2 or W3 according to EHS classification) will be included in La Fe Hospital in Valencia from January 2017 until the recruitment of the entire sample (estimated in December 2018).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old (men and women).
* To give his consent to participation in the study.
* To have surgical prosthetic repair of large incisional hernia (type W2 or W3).
* Patients admitted to the 6th floor, G tower (Unit of Abdominal Wall surgery).

Exclusion Criteria:

* Patients with immediate reintervention of abdominal surgery (less than 30 days from the first surgery).
* Patients after emergency surgery.
* Patients with biological prosthesis.
* Pregnancy and lactation.
* Hepatic cirrhosis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
questionnaire | 1 YEAR
  data about surgical site occurrences

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari La Fe, Valencia, Spain

REFERENCES:
- [Result] Gomoll AH, Lin A, Harris MB. Incisional vacuum-assisted closure therapy. J Orthop Trauma. 2006 Nov-Dec;20(10):705-9. doi: 10.1097/01.bot.0000211159.98239.d2. PMID 17106382
- [Result] Stannard JP, Zane Atkins B, O'Malley D, Singh H, Bernstein B, Fahey M, Masden D, Attinger CE. use of negative pressure therapy on closed surgical incisions: a case series. Wounds. 2009 Aug;21(8):221-8. PMID 25903674
- [Result] Arroyo AA, Casanova PL, Soriano JV, Torra I Bou JE. Open-label clinical trial comparing the clinical and economic effectiveness of using a polyurethane film surgical dressing with gauze surgical dressings in the care of post-operative surgical wounds. Int Wound J. 2015 Jun;12(3):285-92. doi: 10.1111/iwj.12099. Epub 2013 Jun 7. PMID 23742125
- [Result] Colli A, Camara ML. First experience with a new negative pressure incision management system on surgical incisions after cardiac surgery in high risk patients. J Cardiothorac Surg. 2011 Dec 6;6:160. doi: 10.1186/1749-8090-6-160. PMID 22145641
- [Result] Pellino G, Sciaudone G, Candilio G, Campitiello F, Selvaggi F, Canonico S. Effects of a new pocket device for negative pressure wound therapy on surgical wounds of patients affected with Crohn's disease: a pilot trial. Surg Innov. 2014 Apr;21(2):204-12. doi: 10.1177/1553350613496906. Epub 2013 Jul 24. PMID 23883481
- [Result] de Tullio D, Biondin V, Occhionorelli S. When a postsurgical dehiscence becomes a serious problem. Adv Skin Wound Care. 2011 Nov;24(11):503-6. doi: 10.1097/01.ASW.0000407646.05209.e2. PMID 22015748
- [Result] Ingargiola MJ, Daniali LN, Lee ES. Does the application of incisional negative pressure therapy to high-risk wounds prevent surgical site complications? A systematic review. Eplasty. 2013 Sep 20;13:e49. eCollection 2013. PMID 24106562
- [Result] Wilkes RP, Kilpad DV, Zhao Y, Kazala R, McNulty A. Closed incision management with negative pressure wound therapy (CIM): biomechanics. Surg Innov. 2012 Mar;19(1):67-75. doi: 10.1177/1553350611414920. Epub 2011 Aug 25. PMID 21868417
- [Result] Atkins BZ, Wooten MK, Kistler J, Hurley K, Hughes GC, Wolfe WG. Does negative pressure wound therapy have a role in preventing poststernotomy wound complications? Surg Innov. 2009 Jun;16(2):140-6. doi: 10.1177/1553350609334821. Epub 2009 May 21. PMID 19460818
- [Result] Cima R, Dankbar E, Lovely J, Pendlimari R, Aronhalt K, Nehring S, Hyke R, Tyndale D, Rogers J, Quast L; Colorectal Surgical Site Infection Reduction Team. Colorectal surgery surgical site infection reduction program: a national surgical quality improvement program--driven multidisciplinary single-institution experience. J Am Coll Surg. 2013 Jan;216(1):23-33. doi: 10.1016/j.jamcollsurg.2012.09.009. Epub 2012 Nov 2. PMID 23127793
- [Result] Anderson DJ, Kaye KS, Classen D, Arias KM, Podgorny K, Burstin H, Calfee DP, Coffin SE, Dubberke ER, Fraser V, Gerding DN, Griffin FA, Gross P, Klompas M, Lo E, Marschall J, Mermel LA, Nicolle L, Pegues DA, Perl TM, Saint S, Salgado CD, Weinstein RA, Wise R, Yokoe DS. Strategies to prevent surgical site infections in acute care hospitals. Infect Control Hosp Epidemiol. 2008 Oct;29 Suppl 1:S51-61. doi: 10.1086/591064. No abstract available. PMID 18840089
- [Derived] Bueno-Lledo J, Franco-Bernal A, Garcia-Voz-Mediano MT, Torregrosa-Gallud A, Bonafe S. Prophylactic Single-use Negative Pressure Dressing in Closed Surgical Wounds After Incisional Hernia Repair: A Randomized, Controlled Trial. Ann Surg. 2021 Jun 1;273(6):1081-1086. doi: 10.1097/SLA.0000000000004310. PMID 33201116